CLINICAL TRIAL: NCT04610684
Title: Chemotherapy and Atezolizumab for Patients With Extensive Stage Small Cell Lung Cancer (SCLC) With Untreated, Asymptomatic Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Jeffrey Clarke (Other)
Collaborators: Genentech, Inc. (Industry); Duke University (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Clarke, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN19-427
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Small-cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms | interventions — Carboplatin; Etoposide; atezolizumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Treatment Arm (Experimental): 4 cycles of induction treatment with Atezolizumab (1200 mg on Day 1) combined with carboplatin (5-6 AUC on Day 1) and etoposide (80-100 mg/m2 on Days 1-3). After 4 cycles of induction treatment, subjects will receive atezolizumab maintenance 1200 mg on Day 1 of each 3-week cycle.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin 5-6 mg/mL/min AUC will be delivered over 30 - 60 minutes intravenously on Day 1 of each 21 day Cycle after completion of atezolizumab. For 4 cycles.
  Other Names: paraplatin
Drug: Etoposide — Etoposide 80-100 mg/m2 will be delivered over 60 minutes intravenously on Days 1-3 of each 21 day Cycle after completion of carboplatin (Day 1 only). For 4 cycles.
  Other Names: VP-16
Drug: Atezolizumab — Atezolizumab 1200 mg will be delivered over 60 (± 15) minutes intravenously on Day 1 of each 21 day Cycle for 4 cycles then continue as monotherapy maintenance with the same schedule.
  Other Names: Imfinzi

SUMMARY:
This is a single arm, multicenter phase II trial for 60 patients with untreated extensive stage (ES) small cell lung cancer (SCLC) with asymptomatic brain metastases. Subjects will receive 4 cycles of induction treatment with Atezolizumab (1200 mg on Day 1) combined with carboplatin (5-6 AUC on Day 1) and etoposide (80-100 mg/m2 on Days 1-3). Each cycle equals 21 days. After 4 cycles of induction treatment, subjects will receive atezolizumab maintenance 1200 mg on Day 1 of each 3-week cycle. Subjects will receive treatment until disease progression, unacceptable drug-related toxicity, or withdrawal from study for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years with ability and willingness to provide informed consent.
3. ECOG Performance Status of 0-2.
4. Histological confirmation of Small Cell Lung Cancer- Extensive Stage (SCLC) per Veterans Administration Lung Study Group (VALG).
5. At least one untreated asymptomatic brain metastasis that is measurable by RECIST 1.1 that has not been previously irradiated.
6. No prior treatment for metastatic disease. EXCEPTION: A single cycle of chemotherapy (platinum/etoposide) with or without atezolizumab is allowed within 30 days prior to enrollment.
7. Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC.
8. Any prior cancer treatment must be completed at least 6 months prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline. NOTE: a single cycle of chemotherapy (platinum/etoposide) with or without atezolizumab is allowed within 30 days prior to enrollment. NOTE: Extracranial radiation is allowed.
9. A concurrent diagnosis of a separate malignancy is allowed if clinically stable and does not require tumor-directed therapy.
10. Demonstrate adequate organ function as defined in the table below

    * Absolute Neutrophil Count (ANC) ≥ 1.5K/mm3 without GCSF
    * Hemoglobin (Hgb) ≥ 9 g/dL (without transfusion)
    * Lymphocyte Count: ≥ 500/µL
    * Platelet Count: ≥ 100,000/µL without transfusion
    * Calculated creatinine clearance ≥ 50 cc/min OR Serum Cr < 1.5 x institutional ULN
    * Bilirubin ≤ 1.5 × upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) ≤ 2 × ULN without liver metastasis ≤ 5 × ULN with liver metastasis
    * Alanine aminotransferase (ALT) ≤ 2 × ULN without liver metastasis ≤ 5 × ULN with liver metastasis
11. Females of childbearing potential must have a negative serum pregnancy test within 3 days (72 hours) prior to enrollment. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
12. Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception, including at least one method with a failure of < 1% per year, from the time of informed consent until 150 days (5 months) after treatment discontinuation.
13. Negative hepatitis B surface antigen (HBsAg) test, negative total hepatitis B core antibody (HBcAb) test, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test. The HBV DNA test will be performed only for patients who have a positive total HBcAb test. Testing required at screening only if results are not known.
14. Negative hepatitis C virus (HCV) antibody test, or positive HCV antibody test followed by a negative HCV RNA test. The HCV RNA test will be performed only for patients who have a positive HCV antibody test. A positive HCV RNA test is sufficient to diagnose active HCV infection in the absence of an HCV antibody test.
15. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures.

Exclusion Criteria:

1. Known active CNS metastases which are symptomatic. CNS metastases are considered asymptomatic if the patient does not require high dose or escalating corticosteroids or anticonvulsant therapy. Steroid dose must be equivalent to 2 mg of dexamethasone or less daily.

   * Prior steroid use as part of an anti-emetic regimen with chemotherapy is allowed.
   * Patients must be on a stable dose of corticosteroid. No tapering or decreasing dose within 7 days of enrollment.
2. Leptomeningeal disease. Discrete dural-based metastases will be allowed without evidence of leptomeningeal disease.
3. Radiation therapy within 14 days prior to Day 1 of Cycle 1 Day 1. NOTE: Extracranial radiation is allowed.
4. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
5. Known auto-immune conditions requiring systemic immune suppression therapy other than prednisone < 10 mg daily (or equivalent).
6. History of interstitial pneumonitis from any cause.
7. Concurrent severe and/or uncontrolled medical conditions which may compromise participation in the study as assessed by site investigator.
8. Current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment on Cycle 1 Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or chronic obstructive pulmonary disease) are eligible. NOTE: Subjects with active tuberculosis are NOT eligible.
9. Current use of medications specified by the protocol as prohibited for administration in combination with the study drugs. This includes patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to Cycle 1 Day 1. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients who are receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead.
10. History of myocardial infarction, NYHA class II or greater congestive heart failure, or unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to study enrollment.
11. Known history of HIV seropositivity or known acquired immunodeficiency syndrome (AIDS), Testing not required at screening.
12. Requirement for ongoing anticoagulation with heparin, low molecular weight heparin, or other oral anticoagulant (coumadin, DOAC).
13. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). NOTE: Patients with indwelling catheters (e.g., PleurX®) are allowed.
14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
15. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation.
16. History of allergic reactions to carboplatin or etoposide.
17. Intolerance of atezolizumab or other PD-1/PD-L1 axis drug(s), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immune-stimulatory anti-tumor agents.
18. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors
19. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
20. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
21. Treatment with any investigational drug within 28 days prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Clarke, MD, Principal Investigator — Duke University
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - University of Illinois Cancer Center, Chicago, Illinois
  - St. Vincent Anderson Regional Hospital, Anderson, Indiana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Summit Health, Berkeley Heights, New Jersey
  - Duke Cancer Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 : Carboplatin + Etoposide + Atezolizumab: 4 cycles of induction treatment with Atezolizumab (1200 mg on Day 1) combined with carboplatin (5-6 AUC on Day 1) and etoposide (80-100 mg/m2 on Days 1-3). After 4 cycles of induction treatment, subjects will receive atezolizumab maintenance 1200 mg on Day 1 of each 3-week cycle.
  Carboplatin: Carboplatin 5-6 mg/mL/min AUC will be delivered over 30 - 60 minutes intravenously on Day 1 of each 21 day Cycle after completion of atezolizumab. For 4 cycles.
  Etoposide: Etoposide 80-100 mg/m2 will be delivered over 60 minutes intravenously on Days 1-3 of each 21 day Cycle after completion of carboplatin (Day 1 only). For 4 cycles.
  Atezolizumab: Atezolizumab 1200 mg will be delivered over 60 (± 15) minutes intravenously on Day 1 of each 21 day Cycle for 4 cycles then continue as monotherapy maintenance with the same schedule.
Period: Study Treatment
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 2
Period: Follow up
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 3
Completed | 0
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Number analyzed (Participants) | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [61 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
ECOG Performance Status (Baseline) [Count of Participants; unit: Participants] — GRADE ECOG PERFORMANCE STATUS 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 2
    1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Progression Free Survival (iPFS)
Description: Intracranial PFS is defined as the time from Day 1 of treatment until the criteria for intracranial disease progression is met as defined by RANO-BM or death as a result of any cause, whichever comes first. Progression disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From C1D1 until death or up to a maximum of 6 months
Population: This study was terminated early and no analysis was done by the sponsor investigator. Therefore, Intracranial progression free survival status per subject is reported here. If subject progressed per RANO-BM or expired then it is coded as 1, 0 otherwise.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Number analyzed (Participants) | 3
Participants
  Subjects Progressed per RANO-BM | 2
  Subjects did not progress per RANO-BM | 1

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR will include complete response (CR) + partial response (PR) as determined by RECIST 1.1. Complete response is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From C1D1 until death or up to a maximum of 6 months
Population: This study was terminated early and no analysis was done by the sponsor investigator. Therefore, overall response rate status per subject is reported here. If subject recorded any PR/CR per RECIST 1.1 then it is coded as 1, 0 otherwise.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Number analyzed (Participants) | 3
Participants
  Responder | 1
  Non-Responder | 02

3. Secondary Outcome: Extracranial Progression Free Survival (PFS)
Description: Extracranial PFS is defined as the time from Day 1 of treatment until the criteria for extracranial disease progression is met as defined by RECIST 1.1 or death as a result of any cause, whichever comes first.Progression disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From C1D1 until death or up to a maximum of 6 months
Population: This study was terminated early and no analysis was done by the sponsor investigator. Therefore, extracranial progression free survival status per subject is reported here. If subject progressed per RECIST 1.1 or expired then it is coded as 1, 0 otherwise.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Number analyzed (Participants) | 3
Participants
  PFS 1 per RECIST 1.1 | 1
  PFS 0 per RECIST 1.1 | 2

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from Day 1 of treatment until death as a result of any cause.
Time Frame: From C1D1 until death or up to a maximum of 9 months
Population: This study was terminated early and no analysis was done by the sponsor investigator. Therefore, overall survival status per subject is reported here. If subject expired then it is coded as 1, 0 otherwise.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Number analyzed (Participants) | 3
Participants
  Subjects Expired | 2
  Subjects Not Expired | 1

5. Secondary Outcome: Toxicity of Atezolizumab Plus Carboplatin and Etoposide
Description: Toxicity of atezolizumab has been evaluated when administered with carboplatin and etoposide in subjects with untreated SCLC brain metastases.Toxicity will be graded by Common Toxicity Criteria for Adverse Events (CTCAE V5).
Time Frame: From C1D1 until death or up to a maximum of 9 months
Population: This study was terminated early and no analysis was done by the sponsor investigator.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
Number analyzed (Participants) | 3
Participants
  Number of patients had at least one adverse event of any grade | 3
  Number of patients had at least one toxicity grade 3 or greater adverse event | 3
  Number of patients had at least one grade 3 or greater treatment related adverse event | 2
  Number of patients having serious adverse event | 1

ADVERSE EVENTS:
Time Frame: From C1D1 until death or up to a maximum of 9 months
Description: Adverse events will be recorded from the time of consent and for at least 30 days after final protocol treatment or until the start of a new anti-cancer treatment.
  SAEs must be reported during the course of the study within 24 hours of discovery of the event.
Arm/Group | Arm 1 : Carboplatin + Etoposide + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 : Carboplatin + Etoposide + Atezolizumab (N=3)
LUNG INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 : Carboplatin + Etoposide + Atezolizumab (N=3)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 2 (5)
ANXIETY (Psychiatric disorders) | 3 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (3)
DEPRESSION (Psychiatric disorders) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSURIA (Renal and urinary disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 1 (1)
EDEMA TRUNK (General disorders) | 1 (1)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1)
FATIGUE (General disorders) | 3 (3)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (2)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 1 (2)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2)
OBESITY (Metabolism and nutrition disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04610684/Prot_SAP_000.pdf